CLINICAL TRIAL: NCT06599593
Title: Leveraging the Seasonal Malaria Chemoprevention Platform to Address Malaria and Malnutrition
Acronym: INSPIRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Centre de Recherche en Sante de Nouna, Burkina Faso (Other Government); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-42493; 1R21AI182714 (NIH)
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Malaria Incidence; Seasonal Malaria Chemoprevention; Nutrition Assessment; Acute Malnutrition in Childhood; Acute Malnutrition; Integrated Community-based Intervention Package
Keywords: integrated nutritional screening, seasonal malaria chemoprevention, acute malnutrition, malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition-Intervention-SMC Integration (Experimental): In conjunction with SMC administration, CHWs screen children for MUAC. CHW refers children with MUAC <12.5 to the CSPS for MAM/SAM care and to receive all standard nutritional program.
  CHW provides all children ages 6-24 months who do not have acute malnutrition with SQ-LNS (Enov'nutributter; Nutriset; 20 g/day, approximately 100-120 calories).
  Interventions: Dietary Supplement: SQ-LNS; Other: Integrated Nutritional Screening
- Standard of Care Plus SQ-LNS Provision (Active Comparator): Separately from SMC administration, CHWs screen children ages 6-59 months for MUAC as part of their routine program. CHW refers children with MUAC <12.5 to the CSPS for MAM/SAM care and to receive all standard nutritional program.
  CHW provides all children ages 6-24 months who do not have acute malnutrition with SQ-LNS (Enov'nutributter; Nutriset; 20 g/day, approximately 100-120 calories).
  Interventions: Dietary Supplement: SQ-LNS

INTERVENTIONS:
Dietary Supplement: SQ-LNS — CHW provides all children ages 6-24 months who do not have acute malnutrition with SQ-LNS (Enov'nutributter; Nutriset; 20 g/day, approximately 100-120 calories).
Other: Integrated Nutritional Screening — In conjunction with SMC administration, CHWs screen children for MUAC. CHW refers children with MUAC <12.5 to the CSPS for MAM/SAM care and to receive all standard nutritional program.
  Arms: Nutrition-Intervention-SMC Integration

SUMMARY:
In the Sahel, the malaria and malnutrition seasons overlap during the rainy season, from approximately July through October. Malaria transmission increases due to the rain and collection of standing water and malnutrition risk increases because this period is the growing season, leading up to the annual harvest in November. Seasonal malaria chemoprevention (SMC) is an antimalarial intervention that involves monthly distribution of sulfadoxine-pyrimethamine (SP) and amodiaquine (AQ) to children aged 3-59 months during the high malaria transmission season. SMC is distributed to millions of children annually in 13 countries in the Sahel, including Burkina Faso. Although SMC distribution is highly effective against clinical malaria in children, malaria remains a major cause of childhood mortality and morbidity in Burkina Faso. The SMC platform, which involves monthly door-to-door delivery of SP-AQ, is an attractive platform for delivery of additional interventions that may augment child health during this vulnerable season. Malaria and malnutrition co-occur in children and communities, and interventions for one may affect the other. For example, previous work by our group and others has shown that antimalarial treatments may improve weight gain in children with malnutrition. The pilot trial is designed to evaluate how the SMC platform may be leveraged to deliver co-interventions with SMC that may augment its efficacy and reduce the incidence of malaria and malnutrition. It is anticipated that the results of this study will provide formative data for the development and implementation of a full-scale study evaluating the effects of integration of nutritional interventions on the SMC platform. It is anticipated that such a strategy may provide optimal protection for children during the most vulnerable period of the year by delivering interventions monthly on an existing platform that directly reaches millions of children each month.

ELIGIBILITY:
Children will be eligible for inclusion in the trial if they meet all of the following criteria:

* Live in the study community
* Eligible for SMC
* No allergy to peanuts or cow's milk
* Able to orally feed
* Within the eligible age ranges:

  * 6-59 months for passive surveillance
  * 6-24 months for SQ-LNS provision
* Written informed consent from at least one caregiver
* Caregiver is at least 18 years of age

Children will be recruited during normal distribution (via door-to-door delivery) for SMC, which occurs monthly during the malaria season (July through October).

Children ages 3-6 months are eligible for SMC and will be included in nutritional screening and monitoring by default but will not be eligible for SQ-LNS, which is designed for children ages 6-24 months and will not be part of the passive surveillance.

A random sample of children ages 6-24 months during the first month of distribution will be asked to participate in an active surveillance cohort. These children will be followed biweekly for screening for malaria with a rapid diagnostic test and temperature and monthly for dried blood spot and anthropometric measurements.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 438 (Actual)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Clinical malaria incidence | 5 months
  The primary outcome will be the cumulative incidence of clinical malaria, defined as fever (temperature ≥37.5°C) plus a positive RDT, over the course of one SMC season. The primary outcome will be measured in two ways: active case detection and passive detection. For active surveillance, 25 children aged 6-24 months per community (N=500 total) will be randomly selected for biweekly monitoring for malaria using an HRP2-based RDT. For passive surveillance, we will record all uncomplicated malaria diagnoses at primary healthcare facilities.

SECONDARY OUTCOMES:
Alternative malaria Indicators | 5 months
  For children enrolled in active surveillance across both arms, the team will assess the cumulative incidence of malaria parasitemia by RDT with or without fever
Severe malaria | 5 months
  Severe malaria will be diagnosed at participating healthcare facilities and defined as vital organ dysfunction and/or hyperparasitemia. Data on severe malaria cases will be collected by passive surveillance.
All-cause clinic visits. | 5 months
  Primary healthcare data collected via passive surveillance will include all sick child visits during the study period and will include information related to diagnoses and treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Oldenburg, Principal Investigator — University of California, San Francisco
Locations (1):
- Centre de Recherche en Sante de Nouna, Nouna, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
Informed consent documents for the proposed aims will include explicit language informing the participant's caregiver(s) that residual biological specimens, including DNA, may be stored in a biorepository for other scientific investigators. The informed consent documents will contain language permitting secondary use with broad data sharing under controlled access with general use restrictions in GitHub and OSF. Any data shared will be de-identified. Participants will not be contacted or re-consented for future sharing or accessing data through repositories.
  Privacy and confidentiality protections will be consistent with applicable local laws in Burkina Faso. Data will be de-identified by removing all 18 HIPAA identifiers prior to sharing. All data sharing plans will be reviewed and approved by the respective institutional review boards at all participating institutions and will be reviewed during the informed consent process with caregivers. Caregivers may opt out of data sharing, for